CLINICAL TRIAL: NCT04386148
Title: Impact of Obsidian® ASG Autologous Platelet-rich Fibrin Matrix on Anastomotic Healing in Colorectal Surgery
Brief Title: Impact of Obsidian ® ASG on Anastomotic Healing
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Obsidian-20
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Anastomotic Leak Rectum
Keywords: Colorectal surgery; Anastomotic leak; Obisidan
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- laparoscopic colorectal surgery: Patients undergoing laparoscopic colorectal surgery with use of Obsidian ASG® during primary anastomosis.
  Interventions: Procedure: Obsidian ASG®

INTERVENTIONS:
Procedure: Obsidian ASG® — As part of the elective laparoscopic colorectal surgery, an autologous fibrin matrix was used as part of anastomotic technique in conjunction with activated thrombocytes (Obsidian ASG®). During anastomosis, this matrix was applied after resection onto the colorectal tissue surfaces with the aim of triggering tissue regeneration and improved wound healing.

SUMMARY:
The use of regenerative medicine in colorectal surgery constitutes an entirely new therapeutic principle. The aim of this new therapeutic approach is to reduce the anastomotic leak rate and minimise morbidity and mortality. The literature identifies the leak rate for colorectal operations as 3-39%.

DETAILED DESCRIPTION:
Introduction:

The use of regenerative medicine in colorectal surgery constitutes an entirely new therapeutic principle. The aim of this new therapeutic approach is to reduce the anastomotic leak rate and minimise morbidity and mortality. The literature identifies the leak rate for colorectal operations as 3-39%.

Methods:

This is a prospective, multi-centre descriptive study commencing in June 2018. As part of the elective laparoscopic colorectal surgery, an autologous fibrin matrix was used as part of anastomotic technique in conjunction with activated thrombocytes (Obsidian ASG®). During anastomosis, this matrix was applied after resection onto the colorectal tissue surfaces with the aim of triggering tissue regeneration and improved wound healing.

ELIGIBILITY:
Inclusion Criteria:

elective laparoscopic colorectal surgery with a primary anastomosis treatment

Exclusion Criteria:

1. pregnancy
2. Breastfeeding period
3. concomitant disease with the potential for a relevant impairment of the anastomosis durability (leukemia, cirrhosis of the liver, Child Pugh A-C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who undergoing elective laparoscopic colorectal surgery with a primary left-sided anastomosis treatment
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Anastomotic leak rate | 20 days
  Anastomotic leak rate after colorectal surgery with Primary anastomosis

SECONDARY OUTCOMES:
feacal blood | 20 days
  number of Patients with feacal blood after colorectal surgery with Primary anastomosis
fever | 20 days
  number of patients with fever higher than 38°C after colorectal surgery
length of Hospital stay | 20 days
  days spent in Hospital after undergoing colorectal surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for General and Visceral Surgery, Kepler University Clinic Linz, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fraccalvieri D, Biondo S, Saez J, Millan M, Kreisler E, Golda T, Frago R, Miguel B. Management of colorectal anastomotic leakage: differences between salvage and anastomotic takedown. Am J Surg. 2012 Nov;204(5):671-6. doi: 10.1016/j.amjsurg.2010.04.022. Epub 2011 May 19. PMID 21600561
- [Background] Rahbari NN, Weitz J, Hohenberger W, Heald RJ, Moran B, Ulrich A, Holm T, Wong WD, Tiret E, Moriya Y, Laurberg S, den Dulk M, van de Velde C, Buchler MW. Definition and grading of anastomotic leakage following anterior resection of the rectum: a proposal by the International Study Group of Rectal Cancer. Surgery. 2010 Mar;147(3):339-51. doi: 10.1016/j.surg.2009.10.012. Epub 2009 Dec 11. PMID 20004450
- [Background] Buchs NC, Gervaz P, Secic M, Bucher P, Mugnier-Konrad B, Morel P. Incidence, consequences, and risk factors for anastomotic dehiscence after colorectal surgery: a prospective monocentric study. Int J Colorectal Dis. 2008 Mar;23(3):265-70. doi: 10.1007/s00384-007-0399-3. Epub 2007 Nov 22. PMID 18034250